CLINICAL TRIAL: NCT03735225
Title: A Randomized, Double-blind, Placebo-controlled, Doseescalation Trial to Evaluate the Safety and Tolerability of a Single IV Administration of Dasiglucagon and the Bioavailability of Dasiglucagon Following SC Compared to IV Administration in Healthy Subjects
Brief Title: Evaluation of the Safety, Tolerability and Bioavailability of Dasiglucagon Following Subcutaneous (SC) Compared to IV Administration
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Zealand Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZP4207-17144
Record Dates: First submitted 2018-10-10; First posted 2018-11-08 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Hypoglycemia
MeSH Terms: conditions — Hypoglycemia | interventions — dasiglucagon

STUDY DESIGN:
Intervention Model Description: Dose escalation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IV Dasiglucagon (Experimental): Dasiglucagon 0.1, 0.3, 0.6, 1.5 or 2.0 mg administered IV as a single dose
  Interventions: Drug: Dasiglucagon
- SC 0.6 mg Dasiglucagon (Experimental): Dasiglucagon 0.6 mg administered SC as a single dose
  Interventions: Drug: Dasiglucagon
- IV Placebo (Placebo Comparator): Placebo 0.1, 0.3, 0.6, 1.5 or 2.0 mg administered IV as a single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dasiglucagon — Dasiglucagon injection
  Other Names: ZP4207
  Arms: IV Dasiglucagon; SC 0.6 mg Dasiglucagon
Drug: Placebo — Placebo for Dasiglucagon injection
  Other Names: Placebo for Dasiglucagon
  Arms: IV Placebo

SUMMARY:
The purpose of the trial is to characterize the safety and tolerability of dasiglucagon 4 mg/mL following IV administration at increasing doses in healthy volunteers. One cohort of subjects will receive a SC dose of dasiglucagon to characterize the bioavailability of dasiglucagon following SC administration compared to IV administration. Furthermore, the trial aims to assess the potential effect of dasiglucagon on corrected QT interval (QTc) prolongation via a concentrationresponse analysis.

DETAILED DESCRIPTION:
Hypoglycemia in patients with diabetes is defined as episodes of an abnormally low plasma glucose concentration. Hypoglycemia is a common, unpredictable, and potentially dangerous side effect of treatment of diabetes mellitus, especially with insulin or sulfonylureas.

Dasiglucagon (ZP4207) is a stable peptide analog of human glucagon, available in a ready-to-use liquid formulation. Dasiglucagon is in development for the treatment of severe hypoglycemia in patients with diabetes mellitus. Dasiglucagon is a specific and full glucagon receptor agonist designed to mimic the effects of glucagon, having a fast absorption and elimination (minutes).

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities (trial-related activities are any procedures that would not have been performed during normal management of the subject).
* Healthy female or male subjects aged between 18 and 45 years, both inclusive.
* Body weight between 60 and 90 kg, both inclusive.
* Subjects in good health according to age (medical history, physical examination, vital signs, and laboratory assessments), as judged by the investigator.
* Systolic Blood Pressure (SBP) ≥90 mmHg, ≤140 mmHg and Diastolic Blood Pressure (DBP) ≤90 mmHg measured after at least 5 min rest in supine position.
* A pulse rate of ≥50 and ≤90 b/min measured after at least 5 min rest in supine position.
* 12-lead ECG with QTcF < 450 ms, PR < 220 ms and QRS < 110 ms.
* A female subject must meet one of the following criteria:

  * Participant is of childbearing potential and agrees to use one of the accepted contraceptive regimens throughout the entire duration of the trial from screening until the last follow-up visit. An acceptable method of contraception includes one of the following:

    * Total heterosexual sexual abstinence can be used as a method of contraception if this is the participant's preferred lifestyle and the method is established. Periodic sexual abstinence is not an acceptable method of contraception

Single method (use only one method):

* intrauterine device (IUD),
* hormone rod inserted under the skin,
* male partner's sterilization

Double method:

* Hormone contraception A) estrogen and / or progesterone oral contraceptives, B) transdermal patch, C) vaginal ring, D) injection in combination with one of the following: a) vaginal cap with spermicide, b) vaginal sponge (only for women who have never given birth), c) condom, d) female condom
* Participant is of non-childbearing potential, if she is either surgically sterilized (ie, by tubal ligation or removal of ovaries), has undergone complete hysterectomy, or is in a menopausal state (i.e., at least one year without menses).

  * A male subject who is sexually active and has a female partner who is of childbearing potential, must use a condom throughout the entire duration of the trial from screening and until the last follow-up visit.

Condoms MUST be combined with one of the following methods:

* IUD,
* hormone rod inserted under the skin,
* vaginal cap with spermicide,
* vaginal sponge (only for women who have never given birth),
* hormone contraception A) estrogen and / or progesterone oral contraceptives, B) transdermal patch, C) vaginal ring or D) injection

  * Total heterosexual sexual abstinence can be used as a method of contraception if this is the participant's preferred lifestyle and the method is established. Periodic sexual abstinence is not an acceptable method of contraception.

Exclusion Criteria:

* Previous participation in any trial with dasiglucagon. Participation defined as enrolled into trial.
* Known or suspected hypersensitivity to trial product(s) or related products.
* History of severe hypersensitivity to medicines or foods or history of severe medicinal/food induced anaphylactic reaction.
* Receipt of any investigational product within 3 months prior to screening.
* Females who are pregnant according to a positive pregnancy test, are actively attempting to get pregnant, or are lactating.
* Any history or presence of cancer, except adequately treated (as judged by investigator) basal or squamous cell skin cancer or cervical carcinoma in situ.
* A history or presence of any clinically significant respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, hematological, dermatological, venereal, neurological or psychiatric diseases, or other major diseases at the discretion of the investigator.
* Known cardiovascular disease, arthrosclerosis, angina pectoris, or a history of myocardial infarction or coronary arterial bypass graft/percutaneous coronary intervention.
* Clinically significant illness (eg, systemic infection) within 4 weeks before screening, as judged by the investigator.
* Any significant pre-existing medical condition as well as pre-planned procedures or surgeries.
* Positive results for Hepatitis B antigens, Hepatitis C antibodies and/or human immunodeficiency virus (HIV) 1 antigen or HIV1/2 antibodies, at screening.
* Any clinically significant abnormal hematology, biochemistry, or urinalysis screening tests, as judged by the investigator.
* Any of the following abnormal laboratory parameters at screening:

  * alanine aminotransferase (ALT) > upper limit of normal [ULN] + 10%, aspartate aminotransferase (AST) > ULN + 10%,
  * Bilirubin > ULN + 20%
* Renal impairment measured as estimated Glomerular Filtration Rate (eGFR) value of eGFR <90 ml/min/1.73 m2 as defined by Kidney Disease: Improving Global Outcomes (KDIGO) 2012 (14).
* Clinically significant abnormal standard 12-lead ECG after 5 min resting in supine position at screening, as evaluated by the investigator.
* Donation of blood or blood loss of more than 500 mL within 12 weeks prior to screening.
* The use of any non-prescribed systemic medication, except routine vitamins and occasional use of acetylsalicylic acid and paracetamol within 14 days prior to randomization.
* A positive result in the alcohol and/or urine drug screen at the screening visit.
* A history of alcoholism or drug abuse as judged by the investigator
* Smokers (defined as a subject who has been smoking within the last 6 month).
* Subjects with mental incapacity or language barriers that preclude adequate understanding or cooperation, who are unwilling to participate in the trial, or who in the opinion of the investigator should not participate in the trial.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2019-06-24 (Actual); Study Completion 2019-06-24 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | day 1, day 2, day 28
  Change measures from baseline considering nausea, vomiting and diarrhea

SECONDARY OUTCOMES:
Clinical assessment of local tolerability at injection site by physical examination | day-1, day 1, day 2, day 28
  Change measures from baseline in pain, redness, itching, edema, induration/infiltration of skin
Occurrence of anti-drug antibodies (ADA) | day 1 and day 28
  Change measures from baseline
Plasma dasiglucagon profiles following IV administration, Area Under the Curve (AUC) | Pre-dose, 5, 15, 25, 40, 60, 80, 100, 120, 140, 180 and 240 min.
  Change measures from baseline
Plasma dasiglucagon profiles following SC administration, Area Under the Curve (AUC) | Pre-dose, 5, 15, 25, 35, 45, 60, 90, 130, 210 and 300 min.
  Change measures from baseline
Change-from-baseline in ECG for QTcF | From day -1 to day 2 and day 28
  Change measures from baseline
Change-from-baseline in ECG for heart rate (HR) | From day -1 to day 2 and day 28
  Change measures from baseline
Change-from-baseline in ECG for pulse rate (PR) | From day -1 to day 2 and day 28
  Change measures from baseline
Change-from-baseline in ECG for QRS | From day -1 to day 2 and day 28
  Change measures from baseline
Frequency of treatment-emergent T-wave morphology changes and U-waves by Holter monitoring | From day -1 to day 2
  Change measures from baseline

CONTACTS AND LOCATIONS:
Overall Officials: Christina M Sylvest, MSc Pharm, Study Director — Zealand Pharma A/S
Locations (1):
- CRS Clinical Research Services Mannheim GmbH, Mannheim, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tehranchi R, Pettersson J, Melgaard AE, Seitz F, Valeur A, Maarbjerg SJ. Dasiglucagon Effects on QTc in Healthy Volunteers: A Randomized, Placebo-Controlled, Dose-Escalation, Double-Blind Study. Curr Ther Res Clin Exp. 2022 Mar 29;96:100668. doi: 10.1016/j.curtheres.2022.100668. eCollection 2022. PMID 35464292